CLINICAL TRIAL: NCT03205358
Title: A Phase II Study of the Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Healthy Toddlers
Brief Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET54; 2014-004367-20 (EudraCT Number); U1111-1143-8912 (Other: WHO)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; MenACYW Conjugate vaccine; NIMENRIX®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal-vaccine naive toddlers aged 12 to 23 months received a single dose of MenACYW Conjugate vaccine.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 2: NIMENRIX® (Active Comparator): Healthy, meningococcal-vaccine naive toddlers aged 12 to 23 months received a single dose of NIMENRIX® vaccine.
  Interventions: Biological: Meningococcal Polysaccharide groups A, C, W-135 and Y Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular (IM)
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal Polysaccharide groups A, C, W-135 and Y Conjugate Vaccine — 0.5 mL, IM
  Other Names: NIMENRIX®
  Arms: Group 2: NIMENRIX®

SUMMARY:
The purpose of the study was to evaluate the immunogenicity and safety profile of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) Conjugate vaccine when given alone compared to that of the licensed Meningococcal groups A, C, W 135 and Y (NIMENRIX®) Conjugate vaccine.

Observational objectives:

* To evaluate the antibody responses to the antigens (serogroups A, C, Y, and W) present in MenACYW Conjugate vaccine and NIMENRIX® measured by serum bactericidal assay using baby rabbit complement (rSBA) and by serum bactericidal assay using human complement (hSBA)
* To evaluate the antibody responses against tetanus in participants who received MenACYW Conjugate vaccine or NIMENRIX® vaccine
* To evaluate the safety profile of MenACYW Conjugate vaccine and NIMENRIX®

DETAILED DESCRIPTION:
All participants received 1 dose of MenACYW Conjugate vaccine or NIMENRIX® on Day 0 and were evaluated for immunogenicity and safety profile. The duration of each participant's participation in the trial was 30 to 44 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 23 months on the day of the first study visit.
* Born at full term of pregnancy (greater than or equal to [≥] 37 weeks) or with a birth weight ≥2.5 kilogram (kg) (5.5 pounds).
* Inform Consent Form (ICF) had been signed and dated by the parent(s) or other legally acceptable representative (and by an independent witness if required by local regulations).
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and to comply with all trial procedures.
* Covered by health insurance where applicable.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine before the final blood draw except for influenza vaccination, which might be received at least 2 weeks before or after the study vaccine.
* Previous vaccination against meningococcal disease with either the trial vaccine or mono-, or polyvalent polysaccharide or Conjugate meningococcal vaccine containing serogroups A, B, C, W, or Y.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (≥ 2 milligram [mg]/kg/day of prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (i.e., participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Known systemic hypersensitivity to latex.
* Known thrombocytopenia, as reported by the parent/legally acceptable representative.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥38.0 degree Celsius (°C). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2015-08-19 (Actual); Study Completion 2015-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (8):
- Finland (8):
  - Investigational Site Number 005, Espoo
  - Investigational Site Number 006, Helsinki
  - Investigational Site Number 002, Helsinki
  - Investigational Site Number 007, Jarvenpaa
  - Investigational Site Number 008, Oulu
  - Investigational Site Number 001, Pori
  - Investigational Site Number 003, Tampere
  - Investigational Site Number 004, Turku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Vesikari T, Borrow R, Forsten A, Findlow H, Dhingra MS, Jordanov E. Immunogenicity and safety of a quadrivalent meningococcal tetanus toxoid-conjugate vaccine (MenACYW-TT) in healthy toddlers: a Phase II randomized study. Hum Vaccin Immunother. 2020 Jun 2;16(6):1306-1312. doi: 10.1080/21645515.2020.1733869. Epub 2020 Apr 1. PMID 32233959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 31 March 2015 to 17 July 2015 at 8 clinic centers in Finland.
Pre-assignment Details: A total of 188 participants who met all inclusion and none of the exclusion criteria were randomized and vaccinated in the study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy, meningococcal-vaccine naive toddlers aged 12 to 23 months received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) Conjugate vaccine.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: NIMENRIX®
Started | 94 | 94
Completed | 94 | 94
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed on safety analysis set which included those participants who had received at least 1 dose of the study vaccine and had any safety data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: NIMENRIX® | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.44 (0.302) | 1.47 (0.314) | 1.45 (0.308)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 53 | 90
  Male | 57 | 41 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection-Site and Systemic Reaction Following Vaccination With Either MenACYW Conjugate Vaccine or NIMENRIX®
Description: A solicited reaction was defined as an adverse reaction (AR) observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the case report form (CRF) and considered as related to vaccination. Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability. Grade 3 solicited injection site reactions: Tenderness: cries when injected limb was moved or the movement of the injected limb was reduced; Erythema and Swelling: greater than or equal to (≥) 50 millimeter (mm). Grade 3 solicited systemic reactions: Fever: greater than [>] 39.5 degree Celsius (°C); Vomiting: ≥6 episodes per 24 hours or requiring parenteral hydration; crying abnormal: >3 hours; Drowsiness: sleeping most of the time or difficult to wake up; Appetite lost: refuses ≥3 feeds or refuses most feeds; Irritability: inconsolable.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: NIMENRIX®
Number analyzed (Participants) | 94 | 94
Participants
  Any Injection site tenderness | 28 | 31
  Grade 3 Injection site tenderness | 0 | 1
  Any Injection site erythema | 29 | 33
  Grade 3 Injection site erythema | 2 | 1
  Any Injection site swelling | 14 | 17
  Grade 3 Injection site swelling | 1 | 3
  Any Fever | 7 | 4
  Grade 3 Fever | 1 | 0
  Any Vomiting | 4 | 5
  Grade 3 Vomiting | 0 | 0
  Any Abnormal crying | 31 | 37
  Grade 3 Abnormal crying | 1 | 0
  Any Drowsiness | 32 | 26
  Grade 3 Drowsiness | 0 | 0
  Any Loss of appetite | 22 | 34
  Grade 3 Loss of appetite | 1 | 1
  Any Irritability | 49 | 53
  Grade 3 Irritability | 0 | 2

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events (AEs) data were collected from Day 0 up to Day 30 post-vaccination. The solicited reactions (SRs) were collected up to Day 7 after vaccination. Serious AEs were collected throughout the trial (up to 30 days after vaccination).
Description: SR was an AR observed and reported under the conditions (symptom and onset) pre-listed in the case report form (CRF). An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the CRF in terms of diagnosis and/or onset post-vaccination. Analysis was performed on safety analysis set population.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: NIMENRIX®
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/94
Other Adverse Events (participants affected / at risk) | 49/94 | 53/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=94) | Group 2: NIMENRIX® (N=94)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=94) | Group 2: NIMENRIX® (N=94)
Drowsiness (Nervous system disorders) | 32 (32) | 26 (26)
Pyrexia (General disorders) | 2 (2) | 6 (7)
Injection site Tenderness (General disorders) | 28 (28) | 31 (31)
Injection site Erythema (General disorders) | 29 (29) | 33 (33)
Injection site Swelling (General disorders) | 14 (14) | 17 (17)
Fever (General disorders) | 7 (7) | 4 (4)
Abnormal crying (Psychiatric disorders) | 31 (31) | 37 (37)
Irritability (Psychiatric disorders) | 49 (49) | 53 (53)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5)
Loss of appetite (Metabolism and nutrition disorders) | 22 (22) | 34 (34)
Gastroenteritis (Infections and infestations) | 2 (2) | 7 (7)
Nasopharyngitis (Infections and infestations) | 9 (9) | 5 (5)
Otitis media (Infections and infestations) | 4 (4) | 6 (6)
Respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1)
Rhinitis (Infections and infestations) | 7 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.